CLINICAL TRIAL: NCT03383861
Title: Nutrition Status, Bone Mass Density, and Selective Serotonin Reuptake Inhibitors
Brief Title: Nutrition Status, BMD, and SSRIs
Status: Terminated | Type: Observational
Why Stopped: This is not a clinical trial and is only a retrospective chart review. This was inadvertently entered into the system as a clinical trial.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: 174318
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: BMD
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SSRI long-term user: Adults, 655 with an SSRI prescription ≥180 days and identified in the National Health and Nutrition Examination Survey (NHANES) data.
  Interventions: Diagnostic Test: Dual-Energy X-ray Absorptiometry (DXA)
- Non-user: Adults, 12,372 non-users, were identified in the National Health and Nutrition Examination Survey (NHANES) data.
  Interventions: Diagnostic Test: Dual-Energy X-ray Absorptiometry (DXA)

INTERVENTIONS:
Diagnostic Test: Dual-Energy X-ray Absorptiometry (DXA) — BMD t-score derived from DXA scan

SUMMARY:
The association between selective serotonin reuptake inhibitor (SSRI) use and bone mass density (BMD) has been debated. Some have suggested features of depression, which SSRIs are prescribed to treat, may be a cause of decreased BMD, such as poor overall food intake at the time of SSRI use. Our study seeks to determine whether SSRI use in adults is associated with lower than average BMD, and if there is an association between low micronutrient intake, SSRI use, and a low BMD.

ELIGIBILITY:
Inclusion Criteria:

* Included adult NHANES participants are those who participated in the Dual-Energy X-ray Absorptiometry (DXA) femur-neck BMD test and responded in full to the demographic, pharmaceutical, and dietary surveys.

Exclusion Criteria:

* Pregnancy, incomplete survey responses, incomplete DXA results

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NHANES participants
Sampling Method: Probability Sample
Enrollment: 13027 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
BMD t-score | NHANES DXA measurement taken 2005-2014

IPD SHARING:
Plan to Share IPD: Undecided